CLINICAL TRIAL: NCT01353872
Title: Effects of Ingestion of Different Sports Drinks on Fatigue During Playing Tennis
Brief Title: Nutrition Effects on Fatigue During Tennis Playing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lescuyer Laboratory (Industry)
Collaborators: Service de Médecine du Sport et des Explorations Fonctionnelles - CHU G Montpied - Clermont-Ferrand (Unknown); Université Blaise Pascal, Clermont-Ferrand (Other)
Responsible Party: Peltier, Lescuyer Laboratory
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 2010-A00724-35
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Fatigue
Keywords: Fatigue; Tennis; Nutrition; Tournament simulation; Delivery of Health Care
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sports Drinks (Experimental): 3 drinks : Nutrattente (before each match) / Nutraperf (during each match) / Nutrarecup (after each match)
  Interventions: Dietary Supplement: Nutrattente / Nutraperf / Nutrarecup
- Placebo (Placebo Comparator): 3 drinks : Nutrattente placebo (before each match) / Nutraperf placebo(during each match) / Nutrarecup placebo (after each match)
  Interventions: Dietary Supplement: Nutrattente placebo / Nutraperf placebo / Nutrarecup placebo

INTERVENTIONS:
Dietary Supplement: Nutrattente / Nutraperf / Nutrarecup — 500 mL of Nutrattente before each match 500 mL/h of Nutraperf during each match 250 mL of Nutrarecup after each match
  Arms: Sports Drinks
Dietary Supplement: Nutrattente placebo / Nutraperf placebo / Nutrarecup placebo — 500 mL of Nutrattente placebo before each match 500 mL/h of Nutraperf placebo during each match 250 mL of Nutrarecup placebo after each match
  Arms: Placebo

SUMMARY:
The main objective of this study is to investigate the effects of ingestion of different sports drinks (Nutrattente / Nutraperf / Nutrarecup) on fatigue induced by a tennis tournament simulation.

ELIGIBILITY:
Inclusion Criteria:

* About 18 to 35 years (inclusive) Subject has a stable weight for at least three months before the start of the study
* Subject able and willing to comply with the protocol and agreeing to give their consent in writing
* Subject affiliated with a social security scheme
* Subject willing to be included in the national register of volunteers who lend themselves to biomedical research

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
peripheral fatigue measured by surface electromyographic (EMG) signal from the right triceps muscle | 3 matches (1.5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Peltier, PhD, Study Director — Lescuyer Laboratory
Locations (1):
- Sirvent, Aubière, France

REFERENCES:
- [Derived] Brink-Elfegoun T, Ratel S, Lepretre PM, Metz L, Ennequin G, Dore E, Martin V, Bishop D, Aubineau N, Lescuyer JF, Duclos M, Sirvent P, Peltier SL. Effects of sports drinks on the maintenance of physical performance during 3 tennis matches: a randomized controlled study. J Int Soc Sports Nutr. 2014 Sep 2;11:46. doi: 10.1186/s12970-014-0046-7. eCollection 2014. PMID 25302057